CLINICAL TRIAL: NCT07040943
Title: A Clinical Trial Evaluating the Safety, Tolerability, and Preliminary Antitumor Activity of IL - 22BP in Refractory Malignant Solid Tumors.
Brief Title: Clinical Trial of IL - 22BP Safety, Tolerability, and Antitumor Activity in Refractory Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024 (1911)
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Refractory Malignant Solid Tumors; mRNA Vaccine; Interleukin
MeSH Terms: interventions — interleukin-22 receptor; mRNA Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Cohort (Experimental): In this study, three patients were grouped together. Subsequently, doses of 50 μg, 100 μg and 150 μg of the IL-22BP were administered to them respectively. The treatment will be administered by intratumoral injection. Enrolled subjects will receive inoculations of IL22BP injection according to their respective dose groups, which include 5 doses for basic immunization and subsequent personalized treatment. During the basic immunization, the first 4 doses will be given at an interval of 1 week each, and the 5th dose will be inoculated 1 month after the 4th dose.
  Interventions: Biological: IL-22BP

INTERVENTIONS:
Biological: IL-22BP — During the injection of IL-22BP, there were three dose groups, namely 50 μg, 100 μg, and 150 μg of mRNA, with three participants in each dose group, aiming to evaluate the safety and tolerability of the IL-22BP. The treatment will be administered by intratumoral injection. Enrolled subjects will receive inoculations of IL22BP injection according to their respective dose groups, which include 5 doses for basic immunization and subsequent personalized treatment. During the basic immunization, the first 4 doses will be given at an interval of 1 week each, and the 5th dose will be inoculated 1 month after the 4th dose.
  Other Names: mRNA vaccine

SUMMARY:
This study aims to investigate the safety and efficacy of the IL-22BP in patients with refractory malignant solid tumors.

DETAILED DESCRIPTION:
Cancer is a leading global cause of death, with advanced cases posing significant treatment challenges due to low efficacy and severe side effects. Gene therapy, especially mRNA-based immunogene therapy, offers promise. IL-22 promotes tumor progression, and its antagonist, IL-22BP, can inhibit tumor growth.

Patients with refractory, metastatic solid tumors unresponsive to second-line therapy lack viable options. This study aims to establish a novel IL-22BP-based mRNA treatment for advanced cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: aged ≥ 18 years old and ≤ 70 years old;
2. Patients with histopathologically confirmed, refractory to second-line treatment, advanced recurrent/metastatic malignant solid tumors and without standard clinical treatment regimens (such as patients with advanced soft tissue sarcoma, advanced head and neck squamous cell carcinoma, malignant melanoma, etc.);
3. Eastern Cooperative Oncology Group (ECOG) performance status score: 0 - 1;
4. Expected survival time ≥ 3 months;
5. More than 28 days since the last chemotherapy/radiotherapy/surgery;
6. More than 6 weeks since the last use of nitrosoureas or mitomycin C;
7. Main organ functions are in good condition;
8. Sign a written informed consent form.

Exclusion Criteria:

1. Have participated in other drug clinical trials within 4 weeks;
2. The tumor is located close to major blood vessels or the trachea;
3. Patients with uncontrolled cardiac clinical symptoms or diseases, such as heart failure of NYHA class II or above, unstable angina pectoris, having had a myocardial infarction within 1 year, and having clinically significant supraventricular or ventricular arrhythmias that require treatment or intervention.
4. For female subjects: pregnant or lactating women.
5. Patients have active tuberculosis, bacterial or fungal infections (≥ grade 2 of NCI-CTCAE 5.0); have active HIV infection, active HBV infection, or HCV infection.
6. Those with a history of psychotropic drug abuse who are unable to quit or have mental disorders;
7. Subjects have any active autoimmune diseases or a history of autoimmune diseases (such as, but not limited to: uveitis, enteritis, hypophysitis, nephritis, hyperthyroidism, hypothyroidism; subjects with vitiligo or those whose asthma in childhood has been completely relieved and who do not require any intervention in adulthood can be included; subjects with asthma that requires bronchodilators for medical intervention cannot be included).
8. Subjects are currently receiving immunosuppressive treatment.
9. Have a history of drug abuse or known medical, psychological, or social conditions, such as a history of alcoholism or drug use.
10. Known to be allergic, hypersensitive, or intolerant to the studied IL-22BP (including any excipients). Have a severe allergy history to any drugs, foods, or vaccines in the past, such as anaphylactic shock, allergic laryngeal edema, allergic dyspnea, allergic purpura, thrombocytopenic purpura, local allergic necrotizing reaction (Arthus reaction), etc.
11. From the screening period to 12 months after the completion of drug injection, female subjects have pregnancy plans or the partners of male subjects have pregnancy plans.
12. According to the investigator's judgment, there are concomitant diseases that seriously endanger patient safety or affect the patient's completion of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-06-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety | Participation in the whole process of the study. The time window was typically 2 months.
  Evaluate the incidence of dose-limiting toxicity during the treatment with IL-22BP formulation and the number of treatment interruptions due to treatment-related adverse reactions during the first treatment cycle.

SECONDARY OUTCOMES:
Objective Response Rate | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP was injected.The time window was typically 2 months.
  It refers to the proportion of patients whose tumors have shrunk to a certain extent and remained so for a certain period of time. It is a direct indicator to measure the anti-tumor activity of drugs.It is usually calculated as the percentage of the sum of the number of patients with complete response (CR) and partial response (PR) in the total number of patients.
Disease Control Rate | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP was injected.The time window was typically 2 months.
  It refers to the proportion of patients whose tumors have shrunk or remained stable. It reflects the control of tumor growth by treatment, including tumor shrinkage (as involved in ORR) and the situation where the tumor does not progress.It is calculated as the percentage of the sum of the number of patients with complete response (CR), partial response (PR), and stable disease (SD) in the total number of patients.
Time to first complete remission, partial remission on treatment with IL-22BP preparation. | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP was injected.The time window was typically 2 months.
  Complete Response: All target lesions disappear, no new lesions emerge, and tumor markers return to normal. This means that, from the perspective of imaging and relevant examinations, the tumor has completely vanished, and the patient's condition has achieved the most ideal improvement. For example, in the treatment of lymphoma, if enlarged lymph nodes completely disappear as detected by imaging examinations such as PET-CT, and relevant tumor markers in the blood also return to normal, it can be judged as a complete response.
  Partial Response: The sum of the maximum diameters of target lesions is reduced by ≥ 30%, and no new lesions appear. Taking lung cancer as an example, if the sum of the maximum diameters of lung tumors is reduced by more than 30% after treatment and no new tumor lesions are detected, it is in a partial response state. This situation indicates that the tumor responds to the treatment and the patient's condition is under a certain degree of control.
Duration of Response | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP was injected.The time window was typically 2 months.
  It is defined as the time between the first confirmation of complete response, partial response and the first disease progression or death from any cause.
Progression - Free Survival(PFS) | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP was injected. The time window was typically 2 months.
  Defined as the time between first treatment with IL-22BP and first disease progression or death from any cause progression or death from any cause.
Overall Survival(OS) | From the time when the patients were enrolled in the study until one month after the last dose of the IL-22BP was injected. The time window was typically 2 months.
  OS defined as time from first treatment with IL-22BP to death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Department of Radiation Oncology, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Gersten O, Barbieri M. Evaluation of the Cancer Transition Theory in the US, Select European Nations, and Japan by Investigating Mortality of Infectious- and Noninfectious-Related Cancers, 1950-2018. JAMA Netw Open. 2021 Apr 1;4(4):e215322. doi: 10.1001/jamanetworkopen.2021.5322. PMID 33843999
- [Background] Kempski J, Giannou AD, Riecken K, Zhao L, Steglich B, Lucke J, Garcia-Perez L, Karstens KF, Wostemeier A, Nawrocki M, Pelczar P, Witkowski M, Nilsson S, Konczalla L, Shiri AM, Kempska J, Wahib R, Brockmann L, Huber P, Gnirck AC, Turner JE, Zazara DE, Arck PC, Stein A, Simon R, Daubmann A, Meiners J, Perez D, Strowig T, Koni P, Kruglov AA, Sauter G, Izbicki JR, Guse AH, Rosch T, Lohse AW, Flavell RA, Gagliani N, Huber S. IL22BP Mediates the Antitumor Effects of Lymphotoxin Against Colorectal Tumors in Mice and Humans. Gastroenterology. 2020 Oct;159(4):1417-1430.e3. doi: 10.1053/j.gastro.2020.06.033. Epub 2020 Jun 22. PMID 32585307
- [Background] Hou X, Zaks T, Langer R, Dong Y. Lipid nanoparticles for mRNA delivery. Nat Rev Mater. 2021;6(12):1078-1094. doi: 10.1038/s41578-021-00358-0. Epub 2021 Aug 10. PMID 34394960
- [Background] Kiaie SH, Majidi Zolbanin N, Ahmadi A, Bagherifar R, Valizadeh H, Kashanchi F, Jafari R. Recent advances in mRNA-LNP therapeutics: immunological and pharmacological aspects. J Nanobiotechnology. 2022 Jun 14;20(1):276. doi: 10.1186/s12951-022-01478-7. PMID 35701851